CLINICAL TRIAL: NCT05283447
Title: Effectiveness of Manual Therapy in the Treatment of Gastroesophageal Reflux Disease in Patients With Type I Hiatal Hernia
Brief Title: Manual Therapy and Gastroesophageal Reflux Disease in Patients With Hiatal Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escoles Universitaries Gimbernat (Other)
Collaborators: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Ricard Tutusaus, Principal Investigator, Escoles Universitaries Gimbernat
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018308
Record Dates: First submitted 2022-02-18; First posted 2022-03-17 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2022-03

CONDITIONS: Gastroesophageal Reflux
Keywords: Hernia, Hiatal; Osteopathic Medicine; Musculoskeletal Manipulations; Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux; Hernia, Hiatal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Specific manual therapy for GERD and hiatal hernia
  Interventions: Other: Osteopathic Medicine
- Control (Placebo Comparator): Manual therapy unrelated to GERD and hiatal hernia
  Interventions: Other: Control

INTERVENTIONS:
Other: Osteopathic Medicine — The clinical protocol subject to analysis for the intervention group consists of manual approach techniques for the myofascial and viscerofascial structures of the anterior face of the neck, maneuvers for the mediastinal region, techniques for normalizing the tone of the thoracic diaphragm and its pillars, on the peritoneal ligaments, and caudal traction of the stomach for manual correction of hiatal hernia.
  Arms: Intervention
Other: Control — The physiotherapeutic treatment on the control group consists of an approach to the lumbopelvic joint restrictions and a massage on the inframesocolic abdominal region with minimal pressure, which does not affect the activity and position of the stomach.
  Arms: Control

SUMMARY:
Introduction: Gastroesophageal reflux disease (GERD) is highly prevalent in our society. The association between GERD and hiatal hernia has been shown to be etiologically critical in the onset or worsening of these patients' clinic. Pharmacological treatment with proton pump inhibitors (IBPs) and H2 blockers is commonly prescribed and will be followed for many patients for life. The cost of health care and the effects of prolonged consumption of PPIs are questionable, and other therapeutic alternatives are being considered. Only in exceptional cases and in patients with GERD and certain types of hiatal hernia is surgery the treatment of choice. Physiotherapy at the time proposed respiratory and diaphragmatic training as a therapeutic alternative that would improve the function of anti-reflux barriers. Recently, other studies evaluating the effectiveness of manual techniques on the crural diaphragm or osteopathic maneuvers on the cervical and thoracic region have obtained good results in the improvement of the MRGE clinic. In this context, the clinical trial presented specifically treats those with reflux disease associated with a Type I hiatal hernia with manual therapy.

Material and methods: The aim of the clinical study is to evaluate the effects of a clinical intervention protocol on patients with GERD for type I hiatal hernia.

The variables are assessed: GERD impact using the GIS MRG Impact Scale, and the EVA format scale for the Reflux Clinic (IEPT) used by the Surgery Service of the Parc Taulí Hospital in Sabadell . The productivity and quality of life of these patients is also assessed using the QOLRAD reflux and dyspepsia patient quality of life questionnaire.

The randomized, double-blind clinical trial has a sample of 44 patients, divided into an intervention group treated with the protocol under study, and a control group undergoing treatment that does not affect the hernia. hiatus and reflux. A total of three treatment sessions are performed on each subject. The participants answer the different questionnaires, before the start of the treatment and for each session, one week after the treatment and one month later. In the protocol, maneuvers are performed on the epigastric region, thoracic diaphragm, mediastinum and anterior face of the neck.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Gastroesophageal Reflux disease (Vakil et al, 2006)
* Age between 18 and 90 years.
* Patients with GERD due to hiatal hernia type I, without surgical indication.
* Patients with GERD due to hiatal hernia type I, with surgical indication on the waiting list.
* Patients with GERD due to hiatal hernia type I, with surgical contraindication.

Exclusion Criteria:

* That fail to meet inclusion criteria.
* Patients treated with Benzodiazepines (BZD)
* Patients with previous surgical interventions at the abdominal level, especially of supramesocolic structures
* Patients diagnosed with Barrett's esophagus
* Patients with paraesophageal and mixed hiatus hernias
* Diagnosed erosive esophagitis
* Active neoplasm
* Serious psychiatric disorders
* Neuromuscular or neurological injuries
* Aneurysms
* Pregnancy
* Hemophilia or treatment with anticoagulant therapy
* Hypersensitivity of the skin or dermatological diseases in the trunk that prevent the performance of the techniques
* Rejection of manual contact

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Impact of GERD (Gastro-oesophageal Reflux Disease) | 8 weeks
  Using "The Gastro-oesophageal Reflux Disease Impact scale" (GIS).The GIS impact assessment scale consists of 9 items that refer to the frequency during the last week of 5 possible symptoms of GERD, the impact on sleep, food or drink intake, work or activities of daily living and the need to use medications in addition to those prescribed by your doctor (from "daily" to "never" on a 4-point Likert-type scale). The Gis scale score ranges from 1 to 4, the higher the score, the better the patient's condition. The scale was validated in Spanish in 2008. (New, Tafalla et al, 2008).

SECONDARY OUTCOMES:
Impact of GERD (Gastro-oesophageal Reflux Disease) | 8 weeks
  Using the "Gastro-oesophageal Reflux Disease impact assessment scale" used by gastroenterology team of the CSPT (Corporación Sanitaria Parc Taulí), aims to objectify GERD symptoms using a 0-10 range. The symptoms generated exclusively by the Reflux will be chosen: heartburn, regurgitation, cough, aphonia, epigastralgia. The maximum sum of the items on the scale is 50 points, indicating maximum severity. The value 0 points would indicate a minimal impact of the disease.
Quality of life in patients with GERD | 8 weeks
  For the collection of specific data on the quality of life of the patients, the QOLRAD scale will be used, this scale contains 25 items, in which the patient is asked about the effect of gastrointestinal symptoms on quality of life. Establishing the relationship with: emotional well-being, sleep, vitality, food and drink, and physical/social functioning. The patient answers the questionnaire about the frequency of these effects in relation to the last week, using a 7-point Likert scale ranging from "all the time/very much" to "never/not at all". Low scores indicate significant impairment in daily functioning (Kulich KR et al, 2005)

CONTACTS AND LOCATIONS:
Overall Officials: Ricard Tutusaus Homs, MSc, Principal Investigator — EU Gimbernat; Salvador Navarro Soto, PhD, Study Director — Corporación Parc Taulí; Alexis Luna Aufroy, PhD, Study Director — Corporación Parc Taulí; Josep Maria Potau Ginés, Study Director — Universidad de Barcelona
Locations (1):
- Ricard Tutusaus Homs, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The pandemic has delayed the completion of the study and no publication date for the information has been proposed.

REFERENCES:
- [Background] El-Serag HB, Sweet S, Winchester CC, Dent J. Update on the epidemiology of gastro-oesophageal reflux disease: a systematic review. Gut. 2014 Jun;63(6):871-80. doi: 10.1136/gutjnl-2012-304269. Epub 2013 Jul 13. PMID 23853213
- [Background] Vakil N, van Zanten SV, Kahrilas P, Dent J, Jones R; Global Consensus Group. The Montreal definition and classification of gastroesophageal reflux disease: a global evidence-based consensus. Am J Gastroenterol. 2006 Aug;101(8):1900-20; quiz 1943. doi: 10.1111/j.1572-0241.2006.00630.x. PMID 16928254
- [Background] Dean C, Etienne D, Carpentier B, Gielecki J, Tubbs RS, Loukas M. Hiatal hernias. Surg Radiol Anat. 2012 May;34(4):291-9. doi: 10.1007/s00276-011-0904-9. Epub 2011 Nov 22. PMID 22105688
- [Background] Bresadola V, Noce L, Ventroni MG, Vianello V, Intini S, Bresadola F. [Sliding hiatal hernia in patients with gastroesophageal reflux: physiopathology and surgical treatment]. Minerva Chir. 2000 Jun;55(6):415-20. Italian. PMID 11059235
- [Background] Savas N, Dagli U, Sahin B. The effect of hiatal hernia on gastroesophageal reflux disease and influence on proximal and distal esophageal reflux. Dig Dis Sci. 2008 Sep;53(9):2380-6. doi: 10.1007/s10620-007-0158-x. Epub 2008 Jan 17. PMID 18205046
- [Background] Smith RE, Sharma S, Shahjehan RD. Hiatal Hernia. 2024 Jul 17. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK562200/ PMID 32965871
- [Background] Patti MG, Goldberg HI, Arcerito M, Bortolasi L, Tong J, Way LW. Hiatal hernia size affects lower esophageal sphincter function, esophageal acid exposure, and the degree of mucosal injury. Am J Surg. 1996 Jan;171(1):182-6. doi: 10.1016/S0002-9610(99)80096-8. PMID 8554137
- [Background] Gryglewski A, Pena IZ, Tomaszewski KA, Walocha JA. Unsolved questions regarding the role of esophageal hiatus anatomy in the development of esophageal hiatal hernias. Adv Clin Exp Med. 2014 Jul-Aug;23(4):639-44. doi: 10.17219/acem/37247. PMID 25166451
- [Background] von Diemen V, Trindade EN, Trindade MR. Hiatal hernia and gastroesophageal reflux: Study of collagen in the phrenoesophageal ligament. Surg Endosc. 2016 Nov;30(11):5091-5098. doi: 10.1007/s00464-016-4858-1. Epub 2016 Mar 22. PMID 27005292
- [Background] Yu HX, Han CS, Xue JR, Han ZF, Xin H. Esophageal hiatal hernia: risk, diagnosis and management. Expert Rev Gastroenterol Hepatol. 2018 Apr;12(4):319-329. doi: 10.1080/17474124.2018.1441711. Epub 2018 Feb 22. PMID 29451037
- [Background] Katz PO, Gerson LB, Vela MF. Guidelines for the diagnosis and management of gastroesophageal reflux disease. Am J Gastroenterol. 2013 Mar;108(3):308-28; quiz 329. doi: 10.1038/ajg.2012.444. Epub 2013 Feb 19. No abstract available. PMID 23419381
- [Background] Wu AH, Tseng CC, Bernstein L. Hiatal hernia, reflux symptoms, body size, and risk of esophageal and gastric adenocarcinoma. Cancer. 2003 Sep 1;98(5):940-8. doi: 10.1002/cncr.11568. PMID 12942560
- [Background] de Burgos Lunar C, Novo del Castillo S, Llorente Diaz E, Salinero Fort MA. [Study of prescription-indication of proton pump inhibitors]. Rev Clin Esp. 2006 Jun;206(6):266-70. doi: 10.1157/13088585. Spanish. PMID 16762289
- [Background] Aguilera-Castro L, Martin-de-Argila-dePrados C, Albillos-Martinez A. Practical considerations in the management of proton-pump inhibitors. Rev Esp Enferm Dig. 2016 Mar;108(3):145-53. doi: 10.17235/reed.2015.3812/2015. PMID 26666270
- [Background] Lopez-Doriga Bonnardeaux P, Neira Alvarez M, Mansilla Laguia S. [Proton bomb inhibitors: a study of the prescription in a functional recovery unit]. Rev Esp Geriatr Gerontol. 2013 Nov-Dec;48(6):269-71. doi: 10.1016/j.regg.2013.07.004. Epub 2013 Oct 5. Spanish. PMID 24099902
- [Background] de la Coba Ortiz C, Arguelles Arias F, Martin de Argila de Prados C, Judez Gutierrez J, Linares Rodriguez A, Ortega Alonso A, Rodriguez de Santiago E, Rodriguez-Tellez M, Vera Mendoza MI, Aguilera Castro L, Alvarez Sanchez A, Andrade Bellido RJ, Bao Perez F, Castro Fernandez M, Giganto Tome F. Proton-pump inhibitors adverse effects: a review of the evidence and position statement by the Sociedad Espanola de Patologia Digestiva. Rev Esp Enferm Dig. 2016 Apr;108(4):207-24. doi: 10.17235/reed.2016.4232/2016. PMID 27034082
- [Background] Eherer AJ, Netolitzky F, Hogenauer C, Puschnig G, Hinterleitner TA, Scheidl S, Kraxner W, Krejs GJ, Hoffmann KM. Positive effect of abdominal breathing exercise on gastroesophageal reflux disease: a randomized, controlled study. Am J Gastroenterol. 2012 Mar;107(3):372-8. doi: 10.1038/ajg.2011.420. Epub 2011 Dec 6. PMID 22146488
- [Background] Nobre e Souza MA, Lima MJ, Martins GB, Nobre RA, Souza MH, de Oliveira RB, dos Santos AA. Inspiratory muscle training improves antireflux barrier in GERD patients. Am J Physiol Gastrointest Liver Physiol. 2013 Dec;305(11):G862-7. doi: 10.1152/ajpgi.00054.2013. Epub 2013 Oct 10. PMID 24113771
- [Background] Carvalho de Miranda Chaves R, Suesada M, Polisel F, de Sa CC, Navarro-Rodriguez T. Respiratory physiotherapy can increase lower esophageal sphincter pressure in GERD patients. Respir Med. 2012 Dec;106(12):1794-9. doi: 10.1016/j.rmed.2012.08.023. Epub 2012 Sep 29. PMID 23026445
- [Background] Ding ZL, Wang ZF, Sun XH, Ke MY. [Therapeutic mechanism of diaphragm training at different periods in patients with gastroesophageal reflux disease]. Zhonghua Yi Xue Za Zhi. 2013 Oct 29;93(40):3215-9. Chinese. PMID 24405544
- [Background] Sun X, Shang W, Wang Z, Liu X, Fang X, Ke M. Short-term and long-term effect of diaphragm biofeedback training in gastroesophageal reflux disease: an open-label, pilot, randomized trial. Dis Esophagus. 2016 Oct;29(7):829-836. doi: 10.1111/dote.12390. Epub 2015 Jul 30. PMID 26227494
- [Background] Qiu K, Wang J, Chen B, Wang H, Ma C. The effect of breathing exercises on patients with GERD: a meta-analysis. Ann Palliat Med. 2020 Mar;9(2):405-413. doi: 10.21037/apm.2020.02.35. Epub 2020 Mar 17. PMID 32233626
- [Background] Eguaras N, Rodriguez-Lopez ES, Lopez-Dicastillo O, Franco-Sierra MA, Ricard F, Oliva-Pascual-Vaca A. Effects of Osteopathic Visceral Treatment in Patients with Gastroesophageal Reflux: A Randomized Controlled Trial. J Clin Med. 2019 Oct 19;8(10):1738. doi: 10.3390/jcm8101738. PMID 31635110
- [Background] Bitnar P, Stovicek J, Hlava S, Kolar P, Arlt J, Arltova M, Madle K, Busch A, Kobesova A. Manual Cervical Traction and Trunk Stabilization Cause Significant Changes in Upper and Lower Esophageal Sphincter: A Randomized Trial. J Manipulative Physiol Ther. 2021 May;44(4):344-351. doi: 10.1016/j.jmpt.2021.01.004. PMID 34090551
- [Background] Martinez-Hurtado I, Arguisuelas MD, Almela-Notari P, Cortes X, Barrasa-Shaw A, Campos-Gonzalez JC, Lison JF. Effects of diaphragmatic myofascial release on gastroesophageal reflux disease: a preliminary randomized controlled trial. Sci Rep. 2019 May 13;9(1):7273. doi: 10.1038/s41598-019-43799-y. PMID 31086250
- [Background] Jones R, Coyne K, Wiklund I. The gastro-oesophageal reflux disease impact scale: a patient management tool for primary care. Aliment Pharmacol Ther. 2007 Jun 15;25(12):1451-9. doi: 10.1111/j.1365-2036.2007.03343.x. PMID 17539985
- [Background] Nuevo J, Tafalla M, Zapardiel J. [Validation of the Reflux Disease Questionnaire (RDQ) and Gastrointestinal Impact Scale (GIS) in patients with gastroesophageal reflux disease in the Spanish population]. Gastroenterol Hepatol. 2009 Apr;32(4):264-73. doi: 10.1016/j.gastrohep.2008.12.004. Epub 2009 Apr 16. Spanish. PMID 19371971
- [Background] Kulich KR, Pique JM, Vegazo O, Jimenez J, Zapardiel J, Carlsson J, Wiklund I. [Psychometric validation of translation to Spanish of the gastrointestinal symptoms rating scale (GSRS) and quality of life in reflux and dyspepsia (QOLRAD) in patients with gastroesophageal reflux disease]. Rev Clin Esp. 2005 Dec;205(12):588-94. doi: 10.1016/s0014-2565(05)72651-5. Spanish. PMID 16527180
- [Background] Sobrino-Cossio S, Soto-Perez JC, Coss-Adame E, Mateos-Perez G, Teramoto Matsubara O, Tawil J, Vallejo-Soto M, Saez-Rios A, Vargas-Romero JA, Zarate-Guzman AM, Galvis-Garcia ES, Morales-Arambula M, Quiroz-Castro O, Carrasco-Rojas A, Remes-Troche JM. Post-fundoplication symptoms and complications: Diagnostic approach and treatment. Rev Gastroenterol Mex. 2017 Jul-Sep;82(3):234-247. doi: 10.1016/j.rgmx.2016.08.005. Epub 2017 Jan 5. English, Spanish. PMID 28065591
- [Background] Pandolfino JE, Shi G, Curry J, Joehl RJ, Brasseur JG, Kahrilas PJ. Esophagogastric junction distensibility: a factor contributing to sphincter incompetence. Am J Physiol Gastrointest Liver Physiol. 2002 Jun;282(6):G1052-8. doi: 10.1152/ajpgi.00279.2001. PMID 12016131